CLINICAL TRIAL: NCT06325202
Title: Closed Loop and Education for Hypoglycemia Awareness Restoration (CLEAR), Conducted by the Impaired Awareness of Hypoglycemia Consortium (IAHC)
Brief Title: Closed Loop and Education for Hypoglycemia Awareness Restoration
Acronym: CLEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Minnesota (Other); University of Kentucky (Other); University of Pennsylvania (Other); AdventHealth (Other); University of Leicester (Other); University of Sheffield (Other); University of Melbourne (Other); Jaeb Center for Health Research (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Vernon Michael Chinchilli, Distinguished Professor, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020946; 1U01DK135126 (NIH)
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: impaired awareness of hypoglycemia; hybrid closed loop device; continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (11):
- current HCL non-user: HCL x 24 months (Experimental): Hybrid closed loop device over a 24-month period for individuals currently not using a hybrid closed loop device
  Interventions: Device: Omnipod 5 or Medtronic 780G
- current HCL non-user: HCL x 12 months, then HCL x an additional 12 months (Experimental): Hybrid closed loop device over a 12-month period for individuals currently not using a hybrid closed loop device, and then a hybrid closed loop device for an additional 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G
- current HCL non-user: HCL x 12 months, then HCL + HARPdoc x 12 months (Experimental): Hybrid closed loop device over a 12-month period for individuals currently not using a hybrid closed loop device, then a hybrid closed loop device plus HARPdoc education for an additional 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G; Behavioral: HARPdoc Education
- current HCL non-user: Usual Care and My HypoCOMPaSS x 12 months, then HCL x 12 months (Active Comparator): Usual Care and My HypoCOMPaSS education over 12 months for individuals currently not using a hybrid closed loop device, then hybrid closed loop device for 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G; Behavioral: My HypoCOMPaSS Education
- current HCL non-user: Usual Care and My HypoCOMPaSS x 24 months (Active Comparator): Usual Care and My HypoCOMPaSS education over 24 months for individuals currently not using a hybrid closed loop device
  Interventions: Behavioral: My HypoCOMPaSS Education
- current HCL user: HCL x 24 months (Experimental): Hybrid closed loop device over a 24-month period for individuals currently using a hybrid closed loop device
  Interventions: Device: Omnipod 5 or Medtronic 780G
- current HCL user: HCL x 12 months, then HCL x an additional 12 months (Experimental): Hybrid closed loop device over a 12-month period for individuals currently using a hybrid closed loop device, and then a hybrid closed loop device for an additional 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G
- current HCL user: HCL x 12 months, then HCL + HARPdoc x 12 months (Experimental): Hybrid closed loop device over a 12-month period for individuals currently using a hybrid closed loop device, then a hybrid closed loop device plus HARPdoc education for an additional 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G; Behavioral: HARPdoc Education
- current HCL user: HCL and My HypoCOMPaSS x 12 months, then HCL x 12 months (Active Comparator): Hybrid closed loop device and My HypoCOMPaSS education over 12 months for individuals currently using a hybrid closed loop device, then hybrid closed loop device for 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G; Behavioral: My HypoCOMPaSS Education
- current HCL user: HCL + My HypoCOMPaSS x 12 months, then HCL + My HypoCOMPaSS + HARPDOC x 12 months (Active Comparator): Hybrid closed loop device and My HypoCOMPaSS education over 12 months for individuals currently using a hybrid closed loop device, then hybrid closed loop device plus My HypoCOMPaSS eduction + HARPdoc education for 12 months
  Interventions: Device: Omnipod 5 or Medtronic 780G; Behavioral: My HypoCOMPaSS Education; Behavioral: HARPdoc Education
- current HCL user: HCL + My HypoCOMPaSS x 24 months (Experimental): Hybrid closed loop device plus My HypoCOMPaSS education over a 24-month period for individuals currently using a hybrid closed loop device
  Interventions: Device: Omnipod 5 or Medtronic 780G; Behavioral: My HypoCOMPaSS Education

INTERVENTIONS:
Device: Omnipod 5 or Medtronic 780G — Omnipod 5 and Medtronic 780G are hybrid closed loop devices that provide automated insulin delivery.
  Arms: current HCL non-user: HCL x 12 months, then HCL + HARPdoc x 12 months; current HCL non-user: HCL x 12 months, then HCL x an additional 12 months; current HCL non-user: HCL x 24 months; current HCL non-user: Usual Care and My HypoCOMPaSS x 12 months, then HCL x 12 months; current HCL user: HCL + My HypoCOMPaSS x 12 months, then HCL + My HypoCOMPaSS + HARPDOC x 12 months; current HCL user: HCL + My HypoCOMPaSS x 24 months; current HCL user: HCL and My HypoCOMPaSS x 12 months, then HCL x 12 months; current HCL user: HCL x 12 months, then HCL + HARPdoc x 12 months; current HCL user: HCL x 12 months, then HCL x an additional 12 months; current HCL user: HCL x 24 months
Behavioral: My HypoCOMPaSS Education — My HypoCOMPaSS is a brief, standardized psycho-educational program delivered in small groups. Facilitated discussions focus on advocating rigorous avoidance of hypoglycemia while maintaining time in target glycemic range.
  Arms: current HCL non-user: Usual Care and My HypoCOMPaSS x 12 months, then HCL x 12 months; current HCL non-user: Usual Care and My HypoCOMPaSS x 24 months; current HCL user: HCL + My HypoCOMPaSS x 12 months, then HCL + My HypoCOMPaSS + HARPDOC x 12 months; current HCL user: HCL + My HypoCOMPaSS x 24 months; current HCL user: HCL and My HypoCOMPaSS x 12 months, then HCL x 12 months
Behavioral: HARPdoc Education — The HARPdoc program targets cognitions around hypoglycemia that act as barriers to hypoglycemia avoidance and recovery of awareness using motivational and cognitive approaches, delivered by diabetes educators, trained and supported by a clinical psychologist, in small group format.
  Arms: current HCL non-user: HCL x 12 months, then HCL + HARPdoc x 12 months; current HCL user: HCL + My HypoCOMPaSS x 12 months, then HCL + My HypoCOMPaSS + HARPDOC x 12 months; current HCL user: HCL x 12 months, then HCL + HARPdoc x 12 months

SUMMARY:
The purpose of the CLEAR study is to determine the effect on counterregulatory responses (CRR) of intervening (by attempting to strictly avoid hypoglycemia) to improve awareness of hypoglycemic symptoms among adults with type 1 diabetes (T1D) who have impaired awareness of hypoglycemia (IAH). IAH affects 20-25% of adults with T1D, and rises with increasing duration of T1D.

DETAILED DESCRIPTION:
Individuals with IAH exhibit blunted symptomatic and CR hormonal responses to hypoglycemia and, as such, have an impaired ability to respond to hypoglycemia. Thus, rates of severe hypoglycemia are up to 6-fold greater in those affected. Intensive management of T1D is necessary in preventing long-term complications, but can be complicated by recurrent episodes of hypoglycemia which lead to and sustain the CRR deficits of IAH. Technologies such as continuous glucose monitoring (CGM) and hybrid closed-loop (HCL) systems can reduce severe hypoglycemia (and also may reduce IAH) but the ability of technology to reverse impaired CRR (as assessed with experimental hypoglycemia clamp) remains unclear. Behavioral and psycho-educational interventions targeting knowledge/skills gaps, as well as particular cognitions and behaviors driving recurrent hypoglycemia, can also reduce severe hypoglycemia and improve awareness. No studies have compared technology with such behavioral interventions in terms of assessing their impact on IAH or the CRR (as a primary outcome). Unanswered questions include the degree of reduction in hypoglycemia required to restore awareness. Furthermore, participants may respond to different interventions according to their characteristics. For example, it remains unclear whether older individuals benefit from such interventions since they usually are excluded from studies. Therefore, there is an urgent need to determine effective interventions that can reverse IAH in a large representative population of adults with T1D and IAH. The investigators propose to study the effect of specific interventions aimed at restoring

* the CRR (tested via an experimental hypoglycemia clamp procedure)
* hypoglycemia awareness (self-reported via the Towler Questionnaire during the experimental hypoglycemia clamp procedure)

The study will use a Sequential Multiple Assignment Randomized Trial (SMART) design. At baseline, all participants who are HCL naïve will be randomized to HCL or Usual Care (UC) plus brief education (My HypoCOMPaSS) with a follow-up of two years. UC will consist of real-time continuous glucose monitoring (CGM) and insulin delivery via pump or multiple daily injections. Participants who fail to increase their CRR at 12 months will be randomized, or assigned, to a second intervention consisting of a small-group educational program focusing on motivations and unhelpful cognitions acting as barriers to hypoglycemia avoidance (HARPdoc). At baseline, all participants who are HCL non-naïve will be randomized to optimized HCL or HCL plus My HypoCOMPaSS; those with non-responsive CRR at 12 months will be randomized to either continue HCL (on the basis they need a longer period to reverse impaired CRR and total symptomatic responses) or to the HARPdoc intervention. Participants randomized to an HCL device are expected to wear the device continually, as well as a CGM. The My HypoCOMPaSS education requires 4-5 hours of training, whereas, the HARPdoc education requires four training sessions of seven hours each during weeks 1,2,3, and 6.

The specific aims and hypotheses are as follows:

Aim 1: To determine the effect on CRR (epinephrine increase ≥ 125 pg/ml over baseline) and total symptom responses (Towler Questionnaire increase ≥ 20% over baseline) during a hyperinsulinemic-hypoglycemic clamp procedure (glucose < 50 mg/dl) after 12 months of HCL versus Usual Care plus My HypoCOMPaSS Educational Intervention among adults with T1D and IAH who have never used HCL therapy previously.

Hypothesis 1: At 12 months, those allocated to Usual Care plus My HypoCOMPaSS will be more likely to have improved CRR and total symptomatic responses than those allocated to HCL.

Aim 2: To determine the effect on CRR and total symptom responses at 12 months of HCL plus My HypoCOMPaSS versus HCL alone among adults with T1D and IAH who are currently using HCL therapy prior to entering the study.

Hypothesis 2: At 12 months, those allocated to HCL plus My HypoCOMPaSS will be more likely to have improved hypoglycemic awareness and improved CRR than those using HCL alone.

Aim 3: To determine the durability of effect over 24 months of the intervention that improves CRR at 12 months among adults with type 1 diabetes and IAH at baseline.

Hypothesis 3: At 24 months, CRR will improve further among those who had restored CRR at 12 months.

Aim 4. To determine the effect on hypoglycemic awareness (Towler Questionnaire increase ≥ 20% over baseline) and CRR (epinephrine increase ≥ 125 pg/ml over baseline) during a hyperinsulinemic hypoglycemic clamp procedure at 24 months of an in-depth educational program (HARPdoc), initiated throughout months 12-24, among adults with T1D and IAH at baseline, for whom the intervention allocated at baseline did not restore CRR at 12 months.

Hypothesis 4: At 24 months, those allocated to HARPdoc for months 12-24 months will be more likely to have improved hypoglycemic awareness and CRR than those who continue with the therapy allocated at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes
* Gold Score or Clarke Score ≥ 4 (highly associated with IAH)
* Random non-fasting C-peptide < 200 pmol/L
* Diabetes duration ≥ 10 years
* HbA1c < 10.5%
* Total Daily Insulin Dose of < 1 unit/kg
* Ability to read and speak English (because validated non-English versions of the cognitive tests and the educational interventions are not available)

Exclusion Criteria:

* Medical conditions that limit participation in study activities, as determined by the PI (including but not limited to cognitive dysfunction, reduced hearing, reduced vision, cancer under active treatment, untreated angina, organ failure)
* Active alcohol or drug abuse (as defined by DSM criteria of either 1) recurrent use of alcohol/drugs resulting in a failure to fulfill major role obligations at work, school, or home, 2) recurrent alcohol/drug use in situations in which it is physically hazardous, or 3) recurrent alcohol or drug-related legal problems)
* Social determinants of health that limit participation in study activities, as determined by the PI (including but not limited to homelessness, food insecurity, inadequate social support)
* Seizure disorder unrelated to hypoglycemia associated seizures, unless documented seizure-free for >12 months and on a stable regimen of anti-convulsant therapy
* Skin conditions that would preclude the use of a CGM
* Super-physiologic exposure to steroids within one month of enrollment
* eGFR < 45 mL/min/1.73 m2
* History of bariatric surgery that irreversibly alters gut innervation and structure
* Hyper- or hypokalemia (serum potassium >5.5 or <3.5 mmol/L)*
* Hemoglobin < 10 g/dL*
* Medical condition that requires intermittent or continuous use of glucocorticoids at greater than physiological replacement doses
* Pregnancy, plan for pregnancy, or breast feeding
* Abnormal thyroid function tests of clinical significance, as determined by PI*
* Liver transaminases > 3 times the upper limit of normal*
* Hospitalization for mental illness in last year
* History of adrenalectomy

  * At discretion of the PI, laboratory tests may be repeated once. If the participant is not eligible after the second attempt, then the participant. The participant may be screened again.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
epinephrine (pg/ml) | measured during the clamp studies at 0 (baseline), 12, and 24 months
  a change in epinephrine (pg/ml) that exceeds 125 pg/ml between (1) 12 months and baseline, and (2) 24 months and baseline
Towler questionnaire | measured during the clamp studies at 0 (baseline), 12, and 24 months
  the Towler questionnaire consists of 12 questions each on a 0-6 Likert scale; a change in the questionnaire that exceeds 20% between (1) 12 months and baseline, and (2) 24 months and baseline

SECONDARY OUTCOMES:
geometric mean of plasma glucagon | measured during the clamp studies at 0 (baseline), 12, and 24 months
  geometric mean of plasma glucagon
geometric mean of plasma pancreatic polypeptide | measured during the clamp studies at 0 (baseline), 12, and 24 months
  geometric mean of plasma pancreatic polypeptide
geometric mean of plasma free fatty acids | measured during the clamp studies at 0 (baseline), 12, and 24 months
  geometric mean of plasma free fatty acids
glucose infusion rate | measured during the clamp studies at 0 (baseline), 12, and 24 months
  glucose infusion rate
HbA1c | measured during the clamp studies at 0 (baseline), 12, and 24 months
  glycated hemoglobin
% of time with sensor hypoglycemia <70 mg/dL | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  % of time with hypoglycemia <70 mg/dL determined from the continuous glucose monitor (CGM) sensor
% of time with sensor hypoglycemia <54 mg/dL | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  % of time with hypoglycemia <54 mg/dL determined from the continuous glucose monitor (CGM) sensor
number of hypoglycemia events | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  number of hypoglycemia events determined from the continuous glucose monitor (CGM) sensor
% time with sensor glucose in range | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  % time with glucose in range determined from the continuous glucose monitor (CGM) sensor
sensor glucose coefficient of variation | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  sensor glucose coefficient of variation determined from the continuous glucose monitor (CGM) sensor
sensor use as the average numbers of days per week | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  sensor use as the average number of days per week determined from the continuous glucose monitor (CGM) sensor
glycemia risk index | measured during the four weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  glycemia risk index determined from the continuous glucose monitor (CGM) sensor
Trail Making Test - Part B | measured during the clamp studies at 0 (baseline), 12, and 24 months
  amount of time required to complete the Trail Making Test - Part B
Four Choice Reaction Time | measured during the clamp studies at 0 (baseline), 12, and 24 months
  Four Choice Reaction Time, which measures reaction time and motor coordination
sleep duration | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  sleep duration determined from an activity monitor smartwatch
sleep quality | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  sleep quality determined by an activity monitor smartwatch
24-hour step count | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  24-hour step count determined by an activity monitor smartwatch
exercise bouts | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  exercise bouts determined by an activity monitor smartwatch
resting heart rate | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  resting heart rate determined by an activity monitor smartwatch
heart rate during exercise | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  heart rate during exercise determined by an activity monitor smartwatch
heart rate variability | measured during the two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  heart rate variability determined by an activity monitor smartwatch
Hypo-METRICS questionnaire | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Hypo-METRICS questionnaire, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
Hypoglycemic Confidence Scale | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Hypoglycemic Confidence Scale, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia, the range is 0 through 27 and higher scores correspond to higher confidence
Hypoglycemia Fear Survey-II | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Hypoglycemia Fear Survey-II, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
Attitudes to Awareness of Hypoglycaemia | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Attitudes to Awareness of Hypoglycaemia, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
Type 1 Diabetes Distress Scale | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Type 1 Diabetes Distress Scale, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
Diabetes Self-Management Questionnaire | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Diabetes Self-Management Questionnaire, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
Diabetes Management Experiences Questionnaire | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  Diabetes Management Experiences Questionnaire, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
PROMIS Sleep Disturbance - Short Form 8a | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  PROMIS Sleep Disturbance - Short Form 8a
Hospital Anxiety and Depression Scale | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months, the range is 0 through 42 and higher scores correspond to higher anxiety and depression
  Hospital Anxiety and Depression Scale
12-Item Hypoglycemia Impact Profile | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  12-Item Hypoglycemia Impact Profile, a Person-Reported Outcome Measure (PROM) specific to hypoglycemia
EQ-5D-5L | measured two weeks prior to each clamp study at 0 (baseline), 12, and 24 months
  EQ-5D-5L, a quality-of-life scale with 5 dimensions
device-related adverse events | throughout the duration of the 24 months of follow-up
  device-related adverse events
severe hypoglycemic events, self-reported on a CLEAR data collection form | throughout the duration of the 24 months of follow-up
  severe hypoglycemic events, self-reported on a CLEAR data collection form
diabetic ketoacidosis (DKA) events | throughout the duration of the 24 months of follow-up
  diabetic ketoacidosis (DKA) events
number of participants with hospitalizations | throughout the duration of the 24 months of follow-up
  number of participants with hospitalizations
number of participants with emergency room (ER) visits | throughout the duration of the 24 months of follow-up
  number of participants with emergency room (ER) visits
major adverse cardiovascular events (MACE) | throughout the duration of the 24 months of follow-up
  major adverse cardiovascular events (MACE)
all-cause mortality | throughout the duration of the 24 months of follow-up
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Vernon M Chinchilli, PhD, Principal Investigator — Penn State College of Medicine; Elizabeth R Seaquist, MD, Study Chair — University of Minnesota; Simon Heller, MD, Study Chair — University of Sheffield
Locations (8):
- United States (5):
  - University of California, San Diego, La Jolla, California
  - AdventHealth, Orlando, Florida
  - University of Kentucky, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Melbourne, Fitzroy, Victoria, Australia
- United Kingdom (2):
  - University of Leicester, Leicester
  - University of Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The release data sets will be stored at the NIDDK Central Repository.
  The release data sets will de-identified, i.e., they will not contain names, social security numbers, addresses, phone numbers, health care records, and/or similar protected health information. In addition, the release data sets will have an anonymous study ID that is linked to an individual only in the participant records at the Biostatistics Research Center at the Penn State College of Medicine.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The timeline for data sharing from the Impaired Awareness of Hypoglycemia Consortium will meet NIH data sharing requirements, such as one year after the Consortium investigators have published the primary manuscript. The Biostatistics Research Center at the Penn State College of Medicine will make data available after the acceptance for publication of the main findings that address the specific aims of the study.
Access Criteria: Investigators external to the Consortium will be able to request the data from the NIDDK Central Repository. They will be required to show proof of their local IRB approval.
URL: https://repository.niddk.nih.gov/home/